CLINICAL TRIAL: NCT01873729
Title: An Open-Label Study of Naltrexone in Adults With Attention Deficit Hyperactivity Disorder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000696
Record Dates: First submitted 2013-05-06; First posted 2013-06-10 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Naltrexone; Adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Naltrexone (Experimental): Naltrexone
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Adults with ADHD

SUMMARY:
The primary aim of this study is to assess whether naltrexone as a monotherapy is effective in treating Attention Deficit Hyperactivity Disorder (ADHD) in adults. Medications that increase dopamine are often effective in treating ADHD in adults. Since naltrexone is a kappa opioid receptor antagonist, it increases dopamine in the brain.

We predict that naltrexone as a monotherapy will be effective for ADHD symptoms in adults with ADHD.

ELIGIBILITY:
Inclusion Criteria

* Male and female outpatients 18-55 years of age.
* Diagnosis of ADHD, by DSM-IV by clinical evaluation by an expert clinician.
* Subjects treated for anxiety disorders and depression who are on a stable medication regimen for at least one month, and who have a disorder-specific CGI-Severity score ≤ 3 (mildly ill) and who have a score on the Hamilton-Depression and Hamilton-Anxiety rating scales below 15 (mild range).

Exclusion Criteria

* Any clinically unstable psychiatric conditions including any history of psychosis or mania, suicidality, sociopathy, criminality, or delinquency.
* Current (last 3 months) substance use disorders (alcohol or drugs),
* Medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study including cardiovascular disease, current untreated hypertension, history of renal or hepatic impairment, or a condition that will or may require treatment with opioid analgesics.
* Clinically significant abnormal baseline laboratory LFT's, which is defined as LFT's greater than the ULN.
* Mental retardation (IQ < 80).
* Organic brain disorders including delirium, dementia, seizures, stroke, neurosurgery, and head trauma with loss of consciousness.
* Pregnant or nursing females.
* Subjects with current adequate treatment for ADHD.
* Current treatment with medication for ADHD.
* Any other concomitant medication with primarily central nervous system activity other than specified in the protocol (a stable and effective treatment regimen of an SSRI or benzodiazepine is permitted per clinical review.)
* A Clinical Global Impression (CGI) of 7 (among the most extremely ill patients) at the screening visit is exclusionary, and any subject who presents a CGI-S of 7 at any point during the study will be removed from participation.
* Subjects presenting with a CGI-Severity score of 6 (severely ill) at two consecutive visits after week 2 will be dropped from the study (i.e. A subject with a CGI of 6 at his/her week 3 visit and at week 4 visit will be dropped from the study at the week 4 visit). Subjects who are dropped for severe or worsening symptoms after exposure to the study medication will receive free follow up care as described in the detailed protocol and protocol summary.
* Non-English speaking subjects

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Naltrexone
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (3.1)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Adult Investigator Symptom Rating Scale (AISRS) Scores From Baseline
Description: The Adult Investigator Symptom Rating Scale (AISRS) is an 18-item clinician rating scale to evaluate individual ADHD symptoms on a scale of 0 (none) to 3 (severe). The total sum ranges from 0 (no ADHD symptoms) to 54 (extremely severe ADHD symptoms).
Time Frame: Baseline and Six weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Naltrexone: Naltrexone + Methylphenidate Spheroidal Oral Drug Absorption System (MPH-SODAS)
  Naltrexone: Adults with ADHD
Arm/Group | Naltrexone
Number analyzed (Participants) | 2
Units on a scale | -5 (5.7)

2. Secondary Outcome: Clinical Global Impression (CGI)
Description: The Clinical Global Impression (CGI) scale allows the clinician to rate the severity of illness, change over time, and efficacy of medication, taking into account the patient's clinical condition and the severity of side effects. The CGI subscales include the Clinical Global Severity of ADHD (CGI-S) which is scored on a 7 point scale (1=not ill, 7=extremely ill) and the Clinical Global Improvement of ADHD (CGI-I) which is also scored on a 7 point scale (1=very much improved, 7=very much worse). The number of subjects with CGI-Improvement scores less than or equal to 2 (very much improved) at the end of the study is reported.
Time Frame: Six weeks
Measure: Number; unit: Participant
Arm/Group | Naltrexone
Number analyzed (Participants) | 2
Participant | 1

ADVERSE EVENTS:
Arm/Group | Naltrexone
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No